CLINICAL TRIAL: NCT01194635
Title: Molecular Correlates of Response to C225 (Erbitux or Cetuximab) in Combination With Cisplatin and Definitive Radiation in Unresectable Stage IV Squamous Cell Carcinoma of the Head and Neck (E3303): A Phase II Trial of Eastern Cooperative Oncology Group
Brief Title: Biomarkers of Response in Blood and Tumor Tissue Samples From Patients With Unresectable Stage IV Squamous Cell Cancer of the Head and Neck Previously Treated With Cetuximab, Cisplatin, and Radiation Therapy
Status: Completed | Type: Observational
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Other Study IDs: CDR0000683306; ECOG-E3303T1
Record Dates: First submitted 2010-09-02; First posted 2010-09-03 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Head and Neck Cancer
Keywords: stage IV squamous cell carcinoma of the lip and oral cavity; stage IV verrucous carcinoma of the oral cavity; stage IV squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the larynx; stage IV verrucous carcinoma of the larynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — In Situ Hybridization, Fluorescence; Gene Expression Profiling; Polymerase Chain Reaction; Enzyme-Linked Immunosorbent Assay; Immunohistochemistry

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

INTERVENTIONS:
Genetic: fluorescence in situ hybridization
Genetic: gene expression analysis
Genetic: polymerase chain reaction
Genetic: protein analysis
Genetic: protein expression analysis
Other: enzyme-linked immunosorbent assay
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of blood and tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors understand how patients respond to treatment.

PURPOSE: This research study is studying biomarkers of response in blood and tumor tissue samples from patients with unresectable stage IV squamous cell carcinoma of the head and neck previously treated with cetuximab, cisplatin, and radiation therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To expand upon the list of molecular correlates indicated in clinical trial ECOG-E3303, including EGFR expression, EGFR phosphorylation, map kinase, AKT, and STAT3.
* To correlate the status or expression level of each biomarker with clinical outcome (response, progression-free survival, overall survival).

OUTLINE: Archived tumor and blood specimens are analyzed for human papilloma virus and p16 status; EGFR gene amplification; levels of ERCC1, XPF, and c-Met proteins; expression and activation of several signaling pathways including PI3 kinase gene and mTOR; levels of ErbB2, ErbB3, P70S6 kinase, S6 , and Akt; expression of amphiregulin (AR), TGF-alpha (TGF-α), heparin-binding EGF-like growth factor (HB-EGF), EGF, epiregulin and c-Met ligand, and hepatocyte growth factor by fluorescence in situ hybridization (FISH), automated in situ quantitative measurements of protein analysis (AQUA), IHC, PCR, and ELISA.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of squamous cell carcinoma of the head and neck

  * Stage IV disease
  * Unresectable disease
* Treated with cetuximab, cisplatin, and radiotherapy on clinical trial ECOG-E3303
* Archived blood and tumor tissue samples available

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Samples from patients enrolled on E3303 from whom samples were submitted for research
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2010-08-05 (Actual); Primary Completion 2010-09-05 (Actual); Study Completion 2010-09-05 (Actual)

PRIMARY OUTCOMES:
Correlation of biomarkers and clinical outcome | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer R. Grandis, MD, Principal Investigator — University of Pittsburgh